CLINICAL TRIAL: NCT04004624
Title: Physiologically Guided Ablation of Reentry-Vulnerable-Zones for the Treatment of Post-Infarction Ventricular Tachycardia
Brief Title: Physiologically Guided VT Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Cardiovascular Reseach and Innovation (Industry)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PhysioVT1
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: This prospective, multi-center controlled study enrolles patients with infarct-related VT refractory to anti-arrhythmic drugs. The outcome of the study group will be compared to historical control group of patients matched for age, LVEF and VT burden.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Arm (Active Comparator): The left ventricle is mapped during atrial and right or left ventricular pacing (site close to the infarct) at a similar cycle length of 600ms. Radio-frequency ablation is performed selectively in areas of activation slowing (defined as ≤40ms per 5mm while voltage abnormalities and late potentials were not specifically targeted.
  Interventions: Device: Ablation
- Control (No Intervention): Patient who underwent ablation using similar technology and irrigated catheters guided by standard substrate mapping techniques.

INTERVENTIONS:
Device: Ablation — Cardiac Ablation
  Arms: Study Arm

SUMMARY:
The purpose of this study is to determine the efficacy of VT ablation guided by functional evaluation of the substrate to specifically target the reentry-vulnerable zones in patients with infarct-related VT.

DETAILED DESCRIPTION:
Activation mapping of VT is the gold-standard method for description of the reentrant circuit and identification of its isthmus, however this is uncommonly accomplished due to hemodynamic non-tolerance and limited temporal and spatial resolution. Substrate mapping has been developed as an alternative method to identify the isthmus of post-infarction VT during sinus rhythm (SR). However, it has limited specificity to critical VT sites.

Fundamental work in animal models of healed infarction and humans has shown that the VT isthmus corresponds to locations characterized by marked activation slowing during SR. Furthermore, these locations serve as "anchors" for multiple VT morphologies and cycle lengths.

The hypothesis of this study is that activation mapping during SR or pacing can improve the specifically for identifying the critical VT sites.

The aim of this prospective, multi-center controlled study is to evaluate the utility and limitations of functional mapping for guiding ablation of reentry vulnerably zones for long-term control of VT

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. History of myocardial infarction ≥1month before enrolment documented by ECG or cardiac imaging (TTE, SPECT, CMR).
3. Planned for first VT ablation procedure.
4. Patients must have an ICD or a plan for ICD implantation after the ablation.
5. Ability to understand the requirement of the study and to sign an informed consent.

Exclusion Criteria:

1. Patients requiring long-term treatment with class I or class III antiarrhythmic drugs after ablation (for AF).
2. The VT substrate is thought not to be related to coronary disease.
3. Presence of ongoing ischemia that is thought to be the cause of the VT.
4. Contraindication to anticoagulation therapy
5. Stroke within 30 days before enrollment.
6. Life expectancy <1 year for any medical condition.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10-12 (Actual); Primary Completion 2019-09-16 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite of VT recurrence or death | 36 months follow-up

IPD SHARING:
Plan to Share IPD: No